CLINICAL TRIAL: NCT01942018
Title: Per Oral Endoscopic Myotomy (POEM) for Esophagogastric Junction Outflow Obstruction (EGOO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00082967
Record Dates: First submitted 2013-09-05; First posted 2013-09-13 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Esophagogastric Junction Outflow Obstruction
Keywords: esophagogastric junction outflow obstruction; EGOO; Per oral endoscopic myotomy; POEM; Gastroesophageal reflux disease; GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EGOO (Experimental): Patients presenting with symptomatic gastroesophageal junction outflow obstruction (EGOO)who will be treated with Per oral endoscopic myotomy (POEM)
  Interventions: Procedure: POEM

INTERVENTIONS:
Procedure: POEM — Patients will receive Per oral endoscopic myotomy (POEM) for symptomatic gastroesophageal junction outflow obstruction (EGOO)

SUMMARY:
This research is being done to study an endoscopic procedure called "POEM" as a less invasive alternative to surgery in people with esophagogastric junction outlet obstruction (EGOO).

DETAILED DESCRIPTION:
Patients with EGOO have difficulty swallowing and/or chest pain. Previously we were not able to distinguish this disease from achalasia. Achalasia is a disease which is characterized by a progressive difficulty with swallowing. It is caused by failure of relaxation of the lower esophageal sphincter (sphincter between esophagus and stomach) along with an essentially aperistaltic esophageal body.

However, EGOO patients have abnormal lower esophageal sphincter relaxation with some preserved peristaltic activity. Because they have some peristalsis, these patients are not diagnosed with achalasia.

Currently, a new diagnostic method, known as high-resolution manometry (HRM), can identify EGOO patients. EGOO patients usually do not respond well to medical treatment and surgery is required in most cases to reduce the pressure of lower esophageal sphincter muscles. This procedure is called "Heller myotomy".

Recently, a new endoscopic method for reducing lower esophageal sphincter pressure has been developed. This method, per-oral endoscopic myotomy (POEM) is now being performed clinically throughout the world, including Johns Hopkins Hospital. The technique utilizes a flexible endoscope to tunnel beneath the esophageal surface layer and cutting muscle fibers of the lower esophagus and upper stomach. POEM is an alternative to invasive surgery with fewer complications. POEM is performed safely at Johns Hopkins Hospital for achalasia patients. Outcomes of POEM have been excellent with greater than 90% positively responding to endoscopic myotomy. Patients with EGOO are being diagnosed more often due to increased use of HRM. They respond poorly to endoscopic therapies but well to surgical myotomy. POEM is the endoscopic equivalent to surgical intervention and represents a less invasive approach to treating these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive adult patients (18-70 years of age) with symptomatic dysphagia (dysphagia score ≥2) EGOO that is diagnosed by high resolution manometry.
2. Ability to give informed consent.

Exclusion Criteria:

1. Unable to give informed consent
2. Pregnant or breastfeeding women (all female patients if child-bearing age will undergo urine pregnancy testing prior to endoscopy)
3. Acute gastrointestinal bleeding
4. Coagulopathy defined by prothrombin time < 50% of control; partial thromboplastin time (PTT) > 50 sec, or international normalized ratio (INR) > 1.5), on chronic anticoagulation, or platelet count <75,000
5. Inability to tolerate sedated upper endoscopy due to cardio-pulmonary instability or other contraindication to endoscopy
6. Prior esophageal or gastric surgeries
7. Cirrhosis with portal hypertension, varices, and/or ascites
8. Active Esophagitis
9. Hiatal hernia larger than 2cm
10. Barrett's esophagus
11. Eosinophilic esophagitis
12. Esophageal stricture
13. Esophageal malignancy
14. Large esophageal diverticulum
15. Mechanical obstruction to esophageal outflow or infiltrative esophageal or gastric disorders.
16. Prior esophageal Botox injection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05; Primary Completion 2020-04 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Change in dysphagia severity | 2 and 6 months
  Dysphagia will be measured by Dysphagia score and Eckhardt score at 2 and 6 months after the procedure (The Eckhardt score takes into consideration symptoms of dysphagia, chest pain, regurgitation and chest pain)

SECONDARY OUTCOMES:
Resolution in Esophago-gastric junction (EGJ) outflow obstruction by HRM performed 2 months after the procedure | 2 months
Change in participants' quality of life | 2 and 6 months
  Improvement in patient's quality of life as reflected by Short Form-36 questionnaire at 2 and 6 months after the procedure
Complication rate | 2 years
  Complications include any of the following (full thickness perforations, unplanned mucosectomies, immediate and delayed bleeding).
Length of hospital stay | 2 years
Procedural times | 2 years
Post procedural Gastroesophageal reflux disease (GERD) | 2 months
  Frequency of post-procedural GERD as documented by either 24 hr ph/Impedence testing, 48 hr Bravo (performed at 2 months), or esophagogastroduodenoscopy (EGD) with evidence of esophagitis
Time to resume normal diet | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mouen A Khashab, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided